CLINICAL TRIAL: NCT03683719
Title: A Phase 2b, Double-blind, Randomised, 5-arm, Vehicle-controlled, Dose-ranging Trial to Evaluate the Efficacy and Safety of Twice Daily Topical Application of Delgocitinib Cream 1, 3, 8, and 20 mg/g for 16 Weeks in Adult Subjects With Mild to Severe Chronic Hand Eczema
Brief Title: Phase 2b Dose-ranging Trial to Evaluate Delgocitinib Cream 1, 3, 8, and 20 mg/g Compared to Delgocitinib Cream Vehicle Over a 16-week Treatment Period in Adult Subjects With Chronic Hand Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-1273
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hand Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Delgocitinib cream 1 mg/g (Experimental): Delgocitinib cream applied twice daily for 16 weeks.
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 3 mg/g (Experimental): Delgocitinib cream applied twice daily for 16 weeks.
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 8 mg/g (Experimental): Delgocitinib cream applied twice daily for 16 weeks.
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 20 mg/g (Experimental): Delgocitinib cream applied twice daily for 16 weeks.
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream vehicle (Placebo Comparator): Delgocitinib cream vehicle applied twice daily for 16 weeks.
  Interventions: Drug: Delgocitinib cream vehicle

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application.
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 1 mg/g; Delgocitinib cream 20 mg/g; Delgocitinib cream 3 mg/g; Delgocitinib cream 8 mg/g
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Other Names: LEO 124249 cream vehicle
  Arms: Delgocitinib cream vehicle

SUMMARY:
The purpose of this research trial was to test different strengths of a new trial medication, delgocitinib cream 1, 3, 8, and 20 mg/g, and to investigate how treatment with delgocitinib cream affects chronic hand eczema. This was judged by a range of assessments that rate the severity and extent of chronic hand eczema and its symptoms, as well as general health status and quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 years or above.
* Diagnosis of chronic hand eczema defined as hand eczema, which has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as mild to severe according to IGA (i.e., IGA ≥2).
* Recent history (within 1 year before the screening visit) of inadequate response to topical corticosteroid treatment or topical corticosteroid treatment being medically inadvisable.
* Diagnostic patch testing performed within 3 years prior to the screening visit.

Key Exclusion Criteria:

* Concurrent skin diseases on the hands e.g tinnea manuum.
* Active atopic dermatitis in regions other than the hands or psoriasis requiring medical treatment.
* Clinically significant infection (e.g., impetiginised hand eczema) on the hands.
* Systemic treatment with immunosuppressive drugs, immunomodulating drugs, retinoids, or corticosteroids within 4 weeks prior to baseline.
* Psoralen ultraviolet A (PUVA) or ultraviolet B (UVB) therapy on the hands within 4 weeks prior to baseline.
* Receipt of live attenuated vaccines 4 weeks prior to baseline.
* Cutaneously applied treatment with immunomodulators (e.g., phosphodiesterase-4 (PDE-4) inhibitors, pimecrolimus, tacrolimus) or topical corticosteroids on the hands within 2 weeks prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 2 weeks prior to baseline.
* Change in systemic antihistamine therapy within 2 weeks prior to baseline i.e., subjects must not start antihistamine treatment or change the current dosage regime within 2 weeks prior to baseline.
* Other cutaneously applied therapy on the hands (except for the use of subject's own emollients) within 1 week prior to baseline.
* Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 1 week prior to baseline.
* Receipt of any marketed or investigational biologic agents within 6 months or 5 half-lives prior to baseline or until cells count returns to normal, whichever is longer.
* Clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to baseline.
* Tuberculosis requiring treatment within 12 months prior to screening and/or subjects with a positive blood test for tuberculosis at screening.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the subject taking antiretroviral medications.
* Any disorder which is not stable and in the investigator's opinion could affect the safety of the subject, influence the findings of the trial, or impede the subject's ability to complete the trial.
* Positive hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (anti-HCV) serology at screening. Subjects with positive HBsAb may be randomised provided they are hepatitis B vaccinated and have negative HBsAg and HBcAb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (25):
- United States (3):
  - Leo Pharma Investigational Site, Tucson, Arizona
  - Leo Pharma Investigational Site, Hialeah, Florida
  - Leo Pharma Investigational Site, Portland, Oregon
- Denmark (4):
  - Leo Pharma Investigational Site, Aarhus
  - Leo Pharma Investigational Site, Copenhagen
  - Leo Pharma Investigational Site, Hellerup
  - LEO Pharma Investigational Site, Herlev
- Germany (18):
  - Leo Pharma Investigational Site, Berlin
  - Leo Pharma Investigational Site, Bochum
  - Leo Pharma Investigational Site, Bremerhaven
  - Leo Pharma Investigational Site, Dresden
  - Leo Pharma Investigational Site, Düsseldorf
  - Leo Pharma Investigational Site, Gera
  - Leo Pharma Investigational Site, Göttingen
  - Leo Pharma Investigational Site, Jena
  - Leo Pharma Investigational Site, Kiel
  - Leo Pharma Investigational Site, Langenau
  - Leo Pharma Investigational Site, Lübeck
  - Leo Pharma Investigational Site, Mahlow
  - Leo Pharma Investigational Site, Mainz
  - Leo Pharma Investigational Site, Memmingen
  - Leo Pharma Investigational Site, München
  - Leo Pharma Investigational Site, Selters
  - Leo Pharma Investigational Site, Stuttgart
  - Leo Pharma Investigational Site, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buhl T, Bauer A, Ehst BD, Thyssen JP, Hahn-Pedersen J, Hagen BF, Apol ED, Agner T. Health-Related Quality of Life in Chronic Hand Eczema in a Phase 2b Trial of Delgocitinib Cream. Dermatol Ther (Heidelb). 2025 May;15(5):1181-1193. doi: 10.1007/s13555-025-01384-4. Epub 2025 Apr 5. PMID 40186746
- [Derived] Weisshaar E, Yuksel YT, Agner T, Larsen LS, Grant L, Arbuckle R, Jones AM, Fromy P, Balita-Crisostomo CL, Mathiasen NN, Thoning H, Apfelbacher C. Development and Validation of a Patient-Reported Outcome Measure of the Impact of Chronic Hand Eczema on Health-Related Quality of Life: the Hand Eczema Impact Scale (HEIS). Dermatol Ther (Heidelb). 2024 Nov;14(11):3047-3070. doi: 10.1007/s13555-024-01267-0. Epub 2024 Oct 21. PMID 39428453
- [Derived] Molin S, Larsen LS, Joensson P, Oesterdal ML, Arbuckle R, Grant L, Skingley G, Schuttelaar MLA. Development and Psychometric Validation of a Patient-Reported Outcome Measure to Assess the Signs and Symptoms of Chronic Hand Eczema: The Hand Eczema Symptom Diary (HESD). Dermatol Ther (Heidelb). 2024 Mar;14(3):643-669. doi: 10.1007/s13555-024-01114-2. Epub 2024 Mar 15. PMID 38485862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 258 participants from 26 sites in 3 countries (U.S., Denmark, Germany) were randomised in this trial. The first participant was screened on 28-Nov-2018 and the last participant completed the trial on 20-Apr-2020.
Pre-assignment Details: 305 participants were screened for this trial. Of these, 47 participants (15.4%) were screening failures. The main reason for screening failure was failure to meet eligibility criteria (11.8%). The eligibility criterion that was most frequently not met was exclusion criterion 21 (positive HBsAg, HBsAb, HBcAb, or antiHCV serology at screening [3.3%]).
Period: Overall Study
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Started | 52 | 51 | 52 | 53 | 50
Completed | 40 | 38 | 44 | 46 | 36
Not Completed | 12 | 13 | 8 | 7 | 14
Not completed — Lack of Efficacy | 1 | 3 | 4 | 0 | 4
Not completed — Adverse Event | 6 | 6 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 4 | 3 | 5 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1
Not completed — Other personal reasons | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle | Total
Number analyzed (Participants) | 52 | 51 | 52 | 53 | 50 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.6) | 46.1 (14.6) | 47.9 (12.9) | 43.9 (15.1) | 47.8 (16.2) | 46.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 28 | 32 | 34 | 27 | 158
  Male | 15 | 23 | 20 | 19 | 23 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 1 | 3 | 9
  Not Hispanic or Latino | 49 | 51 | 50 | 52 | 47 | 249
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 51 | 51 | 50 | 52 | 50 | 254
  Race: Asian | 1 | 0 | 1 | 1 | 0 | 3
  Race: Other | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 5 | 4 | 21
  Denmark | 12 | 7 | 12 | 11 | 16 | 58
  Germany | 36 | 40 | 36 | 37 | 30 | 179
Baseline IGA-CHE score [Count of Participants; unit: Participants] — IGA-CHE is an instrument used in clinical trials to rate the severity of subject's global disease stage and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    0 - Clear | 0 | 0 | 0 | 0 | 0 | 0
    1 - Almost clear | 0 | 0 | 0 | 0 | 0 | 0
    2 - Mild | 13 | 13 | 11 | 12 | 12 | 61
    3 - Moderate | 29 | 29 | 29 | 31 | 27 | 145
    4 - Severe | 10 | 9 | 12 | 10 | 11 | 52
Baseline HECSI score [Mean (Standard Deviation); unit: units on a scale] — HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs of hand eczema and the extent of the lesions on each of 5 hand areas by use of standard scales. The total HECSI score is based on a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and a 5-point scale rating the affected area(s) ranging from 0 (0% affected area) to 4 (76% to 100% affected area). The lowest HECSI score is 0 and the highest possible is 360. A higher HECSI score is indicating more severe hand eczema.
  units on a scale | 59.0 (48.0) | 52.4 (35.9) | 49.5 (29.3) | 65.7 (58.3) | 52.7 (34.9) | 55.9 (42.8)

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment for Chronic Hand Eczema (IGA-CHE) Score of 0 (Clear) or 1 (Almost Clear) With at Least a 2-step Improvement (IGA-CHE Treatment Success) From Baseline to Week 16.
Description: IGA-CHE is an instrument used in clinical trials to rate the severity of subject's global disease stage and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  The multiple comparison procedure - modelling (MCP-Mod) approach was used to guide dose selection. Cochran-Mantel-Haenszel analysis was used to determine the difference in response rates between the active delgocitinib cream doses and delgocitinib cream vehicle.
Time Frame: Week 0 to Week 16.
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 52 | 51 | 52 | 53 | 50
Participants | 11 | 4 | 19 | 20 | 4
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream 3 mg/g vs Delgocitinib Cream 8 mg/g vs Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; The primary endpoint was evaluated by determining if there was a dose-response relationship between the IGA-CHE response rate at Week 16 and the dose administered, using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed and multiple comparison techniques were used to choose the model(s) most likely to represent the true underlying dose-response curve; Test type: Superiority; p < 0.001, Multiple contrast test — P-values were adjusted for multiple comparisons. Models with an adjusted p-value <0.025 were statistically sign. different from a flat dose-response model. Model: IGA-CHE TS = Treatment + Region + Baseline IGA-CHE. Model selected: Emax model
Statistical Analysis 2: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; The difference in response rates between the active delgocitinib cream doses and delgocitinib cream vehicle was analysed separately for each of the active dose groups using the Cochran-Mantel-Haenszel test stratified by region and disease severity (baseline IGA-CHE score). The null hypothesis of no difference in response rates between the delgocitinib cream active doses and delgocitinib cream vehicle was tested against the 2-sided alternative that there is a difference; Test type: Superiority; p > 0.05, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity. Data at visits following premature discont. of IMP or initiation of rescue medication before Week 16 were considered missing and imputed as non-responders (as were any other missing data); Risk Difference (RD) = 13.29, 95% CI 2-sided [0.34 to 26.24]
Statistical Analysis 3: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Risk Difference (RD) = -0.03, 95% CI 2-sided [-10.44 to 10.39]
Statistical Analysis 4: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Risk Difference (RD) = 28.22, 95% CI 2-sided [13.8 to 42.64]
Statistical Analysis 5: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Risk Difference (RD) = 29.61, 95% CI 2-sided [14.56 to 44.67]

2. Secondary Outcome: Change in Hand Eczema Severity Index (HECSI) From Baseline to Week 16.
Description: HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs of hand eczema and the extent of the lesions on each of 5 hand areas by use of standard scales. The total HECSI score is based on a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and a 5-point scale rating the affected area(s) ranging from 0 (0% affected area) to 4 (76% to 100% affected area). The lowest HECSI score is 0 and the highest possible is 360. A higher HECSI score is indicating more severe hand eczema.
  The multiple comparison procedure - modelling (MCP-Mod) approach was used to guide dose selection. A mixed model for repeated measurements (MMRM) analysis was used to determine the difference in the continuous endpoint between the active delgocitinib cream doses and delgocitinib cream vehicle.
Time Frame: Week 0 to Week 16.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 52 | 51 | 52 | 53 | 50
score on a scale | -39.81 (3.71) | -35.93 (3.77) | -46.69 (3.63) | -41.99 (3.59) | -26.40 (3.80)
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream 3 mg/g vs Delgocitinib Cream 8 mg/g vs Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; The secondary endpoint "Change from baseline to Week 16 in HECSI score" was evaluated by determining if there was a dose-response relationship between the change from baseline in HECSI score at Week 16 and the dose administered, using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed and multiple comparison techniques were used to choose the model(s) most likely to represent the true underlying dose-response curve; Test type: Superiority; p < 0.0001, Multiple contrast test — P-values were adjusted for multiple comparisons. Models with an adj. p-value <0.025 were statistically sign. different from a flat dose-response model. Model: Change = Treatment + Baseline + Region + Baseline IGA-CHE. Model selected: Emax model
Statistical Analysis 2: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; Least Square (LS) Means were calculated using a mixed model for repeated measurements on the post-baseline responses up to Week 16 with an unstructured covariance matrix, Kenward-Roger approximation to estimate denominator degrees of freedom, and the mean modelled as follows: Change from baseline in HECSI = treatment × visit + baseline HECSI × visit + region + baseline IGA-CHE. The primary comparison between each active delgocitinib dose and vehicle was at Week 16; Test type: Superiority; p < 0.01, Mixed Models Analysis — The statistical test was not controlled for multiplicity. Data at visits following premature discont. of IMP or initiation of rescue med. before Week 16 were considered missing and imputed with MMRM predicted values (as were any other missing data); Mean Difference (Net) = -13.41, 95% CI 2-sided [-22.82 to -4.01]
Statistical Analysis 3: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = -9.53, 95% CI 2-sided [-19.04 to -0.02]
Statistical Analysis 4: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = -20.29, 95% CI 2-sided [-29.56 to -11.02]
Statistical Analysis 5: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = -15.59, 95% CI 2-sided [-24.82 to -6.36]

3. Secondary Outcome: Time to IGA-CHE Treatment Success.
Description: Time to IGA-CHE treatment success response is defined as the time from baseline to first assessment of an IGA-CHE score of 0 (clear) or 1 (almost clear) with at least a 2-step improvement.
Time Frame: Week 0 to Week 16.
Population: FAS
Measure: Number; unit: days, median
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 52 | 51 | 52 | 53 | 50
days, median | NA — The median time to achieve success in IGA-CHE was not estimable, as fewer participants (less than 50 percent) reached success in IGA-CHE. | NA — The median time to achieve success in IGA-CHE was not estimable, as fewer participants (less than 50 percent) reached success in IGA-CHE. | 82 | 98 | NA — The median time to achieve success in IGA-CHE was not estimable, as fewer participants (less than 50 percent) reached success in IGA-CHE.
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; Time to IGA-CHE TS was defined as the time from the date of the first IMP application to first assessment of IGA-CHE TS. Subjects without baseline observation were censored at the date of the first IMP application. Subjects with baseline observation not achieving IGA-CHE TS during the treatment period were censored at the date of the last visit with a valid post-baseline assessment on or prior to the date of discontinuation of IMP or initiation of rescue medication, whichever occurred first; Test type: Other — Treatment groups were compared using a 2-sided log-rank test stratified by region and baseline IGA-CHE score. An event was defined as the first time achieving IGA-CHE TS; p < 0.05, Log Rank — IGA-CHE TS was reached in less than 50% of participants, therefore the median time was not estimable. The statistical test was not controlled for multiplicity
Statistical Analysis 2: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p > 0.1, Log Rank — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < 0.0001, Log Rank — The statistical test was not controlled for multiplicity
Statistical Analysis 4: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < 0.01, Log Rank — The statistical test was not controlled for multiplicity

ADVERSE EVENTS:
Time Frame: 18 weeks (from first application of IMP up until the last visit (safety follow-up visit))
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/52 | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 2/51 | 1/52 | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 20/52 | 25/51 | 25/52 | 26/53 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 1 mg/g (N=52) | Delgocitinib Cream 3 mg/g (N=51) | Delgocitinib Cream 8 mg/g (N=52) | Delgocitinib Cream 20 mg/g (N=53) | Delgocitinib Cream Vehicle (N=50)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 1 mg/g (N=52) | Delgocitinib Cream 3 mg/g (N=51) | Delgocitinib Cream 8 mg/g (N=52) | Delgocitinib Cream 20 mg/g (N=53) | Delgocitinib Cream Vehicle (N=50)
Nasopharyngitis (Infections and infestations) | 9 (11) | 15 (22) | 15 (16) | 14 (20) | 20 (20)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5) | 3 (7) | 6 (7) | 8 (9)
Headache (Nervous system disorders) | 2 (2) | 2 (4) | 6 (7) | 4 (5) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. After such publication is made public, or if no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03683719/Prot_SAP_000.pdf